CLINICAL TRIAL: NCT06493006
Title: Impact of Physically Active Versus Passive Way to Work on Physical and Mental Aspects of Health in Members at Hannover Universities: an Observational Study
Brief Title: Promoting Sustainable and Active Mobility Among Employees and Students
Acronym: DiNaMo-active
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Gottfried Wilhelm Leibniz Universität Hannover (Other); Hochschule Hannover (Other); Leibniz Information Centre for Science and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01UV2301B
Record Dates: First submitted 2024-06-26; First posted 2024-07-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Mobility on the Way to Work and Health-related Outcomes
Keywords: commuting to work; active mobility; heart rate variability; sustainable universities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long-term group: University members who use mainly one transport mode to get to the work place
- Short-term group: University members who alternate their transport habits between physically active and passive commuting

SUMMARY:
The aim of the study is to assess health data (heart rate variability, blood pressure, blood glucose, particulate matter pollution) and travel characteristics (length, duration and type of commute) on the way to and from work from members of the universities in Hannover (Germany).

DETAILED DESCRIPTION:
Active mobility, (i.e. moving around using the own physical strength) has positive sustainability effects. The physically active way to and from college is a great untapped resources for health promotion. The aim of this sub-project is to examine the way to university in order to assess its effect on individual health depending on the means of transport.

In order to determine the status quo and changes in mobility behavior the investigators will use movement trajectories using smartphone apps or inexpensive trackers in a larger cohort, as well as more specified health measures including overweight status, blood pressure, blood glucose concentration, lack of exercise, particulate matter and risk of accidents in a smaller sub-cohort.

By linking this data with the personal characteristics surveyed in other sub-projects, an evaluation of the individual health status and the expected health benefits depending on the route to work can be created. This represents the database for identifying certain groups of people or status groups who could particularly benefit from targeted promotion of an active commute.

ELIGIBILITY:
Inclusion Criteria:

* living within 50km around the workplace

Exclusion Criteria:

* current participation in another interventional study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees and Students of Hannover Medical School, Leibniz University Hannover, University of Applied Sciences and Arts Hannover, and the Leibniz Information Centre for Science and Technology (all Lower Saxony, Germany)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 24 hours on two separate days for the short-term subgroup, and 7 consecutive days for the long-term subgroup
  HRV measured by a wearable activity tracker

SECONDARY OUTCOMES:
Blood glucose concentration | 24 hours on two separate days for the short-term subgroup
  Intraindividual difference in blood glucose concentration between active and passive commuting as assessed with continuous blood glucose monitoring (Freestyle Libre 3)
Work-Ability-Index | Once at baseline for both study subgroups
  Interindividual difference between work ability as assessed with the Work-Ability-Index-Questionnaire.
  By adding up the points obtained from the questionnaire, scores can range from 7 to 49 points. The lower the score, the greater the discrepancy between the job demands placed on the respondent and their individual ability to cope with them.
24 hour blood pressure | 24 hours on two separate days for the short-term subgroup
  Intraindividual difference in 24 hour arterial blood pressure between active and passive commuting as assessed with 24 hour systolic and diastolic blood pressure monitoring (Boso TM-2450)
Daily moderate to vigorous physical activity (MVPA) duration | 7 consecutive days for the long-term subgroup
  Interindividual difference in MVPA as assessed with a wearable activity tracker (Garmin Smartwatch Forerunner 55)
Health-related quality of life | Once at baseline for both study subgroups
  Interindividual difference between health-related quality of life as assessed with the Short Form 36 questionnaire. The possible score ranges from 0 to 100 points, with 0 points representing the greatest health impairment, while 100 points indicate no health impairment.
Particulate matter | 24 hours on two separate days for the short-term subgroup
  Intraindividual difference in particulate matter concentration between active and passive commuting as assessed with a particulate matter measuring module

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Tegtbur, Prof. Dr., Study Director — Hannover Medical School, Clinic of Rehabilitation and Sports Medicine
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beyer M, Boyen J, Wussow-Hampel S, Stein L, Schmidt LS, Tegtbur U, Haufe S. Role of commuting characteristics on physical and mental health among members at university institutions (DiNaMo-active): a protocol for an observational study. BMJ Open Sport Exerc Med. 2025 Jun 19;11(2):e002665. doi: 10.1136/bmjsem-2025-002665. eCollection 2025. PMID 40546747